CLINICAL TRIAL: NCT06288490
Title: A Single Arm Study Comparing Amorphous Calcium Carbonate (ACC) Supplement Versus Commercially Available Crystalline Calcium Supplements (CCS) in the Management of Hypoparathyroidism
Brief Title: A Single Arm Study Comparing ACC Supplement to CCS in Management of Hypoparathyroidism
Acronym: AMCS009
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: moving to phase II-III
Sponsor: Amorphical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCS-009
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Intervention Model Description: Proof of concept: treatment with smaller doses of elemental calcium from ACC compared to CCS can maintain target serum calcium (corrected for albumin) values (7.0-10.0 mg/dL)
Oversight: Data Monitoring Committee: No

ARMS (1):
- amorphous calcium carbonate (Experimental): Ten (10) subjects previously diagnosed and chronically treated for primary hypoparathyroidism will be enrolled. The daily CCS intake will be gradually replaced by reduced amount of elemental calcium from ACC. Five (5) subjects will consume the ACC before having a meal and the other five (5) subjects will consume the ACC after having a meal. The safety and the efficacy of the treatment will be closely monitored throughout this phase.
  Interventions: Dietary Supplement: amorphous calcium carbonate

INTERVENTIONS:
Dietary Supplement: amorphous calcium carbonate
  Other Names: ACC

SUMMARY:
Primary objective:

Phase I Proof of concept: treatment with smaller doses of elemental calcium from ACC compared to CCS can maintain target serum calcium (corrected for albumin) values (7.0-10.0 mg/dL).

Phase II To test the hypothesis that treatment with smaller doses of elemental calcium from ACC compared to CCS can maintain target serum calcium (corrected for albumin) values (7.0-10.0 mg/dL).

Secondary objectives:

Phase I

* ACC dose selection - to confirm the conversion factor of ACC from CCS
* To determine the effect of food on ACC absorption

Phase II

* To test the hypothesis that treatment with smaller doses of elemental calcium from ACC compared to CCS will not cause an increase in hypercalciuria in patients with hypoparathyroidism
* To test the hypothesis that smaller doses of elemental calcium from ACC can reduce the side effects related with high calcium consumption.

Amorphical has a strong basis to believe that the ACC product is better absorbed compared to the commercially available CCS products and therefore, can maintain desirable target albumin corrected calcium values in serum (CA) with smaller doses of elemental calcium from ACC. As results, the burden of taking high doses of calcium supplementation along with the side effects of the standard therapy (gastrointestinal discomfort and hypercalciuria) will be reduced.

Testing serum CA and urine calcium values in subjects with hypoparathyroidism may provide a straightforward method to test this hypothesis.

The study is designed to be conducted with extra precaution in order to avoid disturbing the fragile balance between CA levels in serum and calcium levels urine. The crossover design of phase II of the study allows a more accurate and reliable comparison of results attributable to the specific treatment within the same individual. In addition, the subjects will continue consuming all their routine medication throughout the trial. The subjects in the control arm will consume their routine calcium supplement doses thus, will be treated with a standard of care.

DETAILED DESCRIPTION:
Eligible subjects will be treated as follows:

Phase I Ten (10) subjects previously diagnosed and chronically treated for primary hypoparathyroidism will be enrolled. The daily CCS intake will be gradually replaced by reduced amount of elemental calcium from ACC. Five (5) subjects will consume the ACC before having a meal and the other five (5) subjects will consume the ACC after having a meal. The safety and the efficacy of the treatment will be closely monitored throughout this phase.

The absorption of ACC will be evaluated using weekly serum calcium corrected for albumin (CA) value tests. Excretion of calcium in urine will be tested at screening and at the end of phase I.

I-Day -21 (+/-17) Screening: Subjects with a diagnosed primary hypoparathyroidism (see section 4.1 for definitions), and who are treated with calcium and vitamin D supplementation at least 1 year prior to the beginning of the study and are without major renal or hepatic disease, will be invited to the Clinical Research Center. At the clinic, subjects will be interviewed, their medical history and their current medication will be documented and they will sign an informed consent form (ICF). Subjects will be referred to perform blood tests for serum calcium, P, creatinine and albumin levels. Calculation of albumin corrected calcium (CA) will be performed. Subjects will be instructed to perform 24 hour urine collection for Ca, P and creatinine. Subjects will be asked to fill out a food and medication diary for 3 consecutive days to evaluate their daily dietary calcium intake. Women of childbearing age will undergo a urine pregnancy test. Eligible subjects, complying with all inclusion criteria and having none of the exclusion criteria will be enrolled to the study.

Subjects will be informed by phone or on site whether they are eligible to enter the study.

I-Day 0: Eligible subjects will arrive at the Clinical Research Center where they will be asked about any changes in their medical condition since their last visit. Blood tests will be performed to define serum calcium, P and albumin baseline values. Calculation CA at baseline will be performed.

Subjects will receive a pack of ACC tablets, each tablet containing 50, 100 or 200 mg elemental calcium (according to the daily total amount of calcium supplementation, 14 day supply + 5 spare tablets). The replacement of CCS with ACC will be calculated according to the following formula:

NTDC = ITDC - [0.1×ITDC (mg CCS)] + [0.05×ITDC (mg ACC)]

*ITDC - Initial total daily calcium intake (mg)

**NTDC - New total daily calcium intake (mg)

10% (in mg) out of the initial total daily intake of elemental calcium will be replaced by 5% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake). The daily intake of vitamin D will remain the same.

The calculation for the number of tablets per day will be performed specifically for each subject (according to the daily dosage of calcium supplementation) by the doctor.

Subjects will be instructed to take XXX ACC tablets a day, according to their individual calculated NTDC:

1. Five subjects will be instructed to take XXX tablets in the morning after a meal, XXX in midday after a meal and XXX in the evening after a meal.
2. Five subjects will be instructed to take XXX tablets in the morning before having a meal, XXX in midday before having a meal and XXX in the evening before having a meal.

Subjects will be instructed to continue their routine medications consumption during the trial.

I-Day 3 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). If CA values are within the desired target range (7.0-10.0 mg/dl), subjects will continue to take the calcium doses that were instructed on I-day 0. If CA values are below 7.0 mg/dl or above 10.0 mg/dl, changes to the calcium intake will be made, according to the doctor's decision.

I-Day 7 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed:

1. Conversion factor 0.5:

   If CA = baseline, then 20% (in mg, calculated out of the initial total daily intake) of elemental calcium will be replaced by 10% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

   NTDC = ITDC - [0.2×ITDC (mg CCS)] + [0.1×ITDC (mg ACC)]
2. Conversion factor 0.75:

   If CA < baseline, then 10% (in mg, calculated out of the initial total daily intake) of elemental calcium will be replaced by 7.5% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

   NTDC = ITDC - [0.1×ITDC (mg CCS)] + [0.075×ITDC (mg ACC)] CA <7.00 mg/dl will enforce end of treatment.
3. Conversion factor 0.25:

If CA > baseline, then 10% (in mg, calculated out of the initial total daily intake) of elemental calcium will be replaced by 2.5% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

NTDC = ITDC - [0.1×ITDC (mg CCS)] + [0.025×ITDC (mg ACC)] Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression). Subjects will receive instructions regarding the new doses of ACC and will be reminded to take XXX tablets a day (according to their individual calculated NTDC), XXX in the morning, XXX in midday and XXX in the evening, before or after a meal (based on their initial assignment). Subjects will be reminded to continue their routine medications consumption during the trial.

I-Day 10 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). If CA levels are within the desired target range (7.0-10.0 mg/dl), subjects will continue to take the calcium doses that were instructed on I-day 7. If CA levels are below 7.0 mg/dl or above 10.0 mg/dl, changes to the calcium intake will be made, according to the doctor's decision.

I-Day 14 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). If none of the conversion formulas (a-c, I-Day 7) resulted in serum calcium values within the desired target range (7.0-10.0 mg/dL), the study will be terminated.

Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

50% of the initial daily supplementation of CCS will be replaced by ACC based on the conversion factor found in I-day 7 (formulas a-c):

1. Conversion factor 0.5: 50% (in mg, calculated out of the initial total daily intake) of elemental calcium will be replaced by 25% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

   NTDC = ITDC - [0.5×ITDC (mg CCS)] + [0.25×ITDC (mg ACC)]
2. Conversion factor 0.75: 50% (in mg, calculated out of the initial total daily intake) of elemental calcium will be replaced by 37.5% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

   NTDC = ITDC - [0.5×ITDC (mg CCS)] + [0.375×ITDC (mg ACC)]
3. Conversion factor 0.25: 50% (in mg, calculated out of the initial total daily intake) of elemental calcium will be replaced by 12.5% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

NTDC = ITDC - [0.5×ITDC (mg CCS)] + [0.125×ITDC (mg ACC)] Subjects will receive a pack of ACC tablets, each tablet containing 50, 100 or 200 mg elemental calcium (according to their individual calculated NTDC, 14 day supply + 5 spare tablets). Subjects will receive instructions regarding the new doses of ACC and will be reminded to take XXX capsules a day, XXX in the morning, XXX in midday and XXX in the evening, before or after a meal (based on their initial assignment). Subjects will be reminded to continue their routine medications consumption during the trial.

I-Day 21 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression). If CA levels are below 7.0 mg/dl, or above 10.0 mg/dl, subject will be excluded from the study (based on the doctor's decision). If CA levels are within the desired target range (7.0-10.0 mg/dL), a complete replacement of the daily supplementation of CCS with ACC will be performed, based on the conversion factor found in I-day 7 (formulas a-c):

1. Conversion factor 0.5: 100% (in mg) of the elemental calcium initial total daily intake will be replaced by 50% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

   NTDC = ITDC - [ITDC (mg CCS)] + [0.5×ITDC (mg ACC)]
2. Conversion factor 0.75: 100% (in mg) of the elemental calcium initial total daily intake will be replaced by 75% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

   NTDC = ITDC - [ITDC (mg CCS)] + [0. 75×ITDC (mg ACC)]
3. Conversion factor 0.25: 100% (in mg) of the elemental calcium initial total daily intake will be replaced by 25% of elemental calcium from ACC (in mg, calculated out of the initial total daily intake).

NTDC = ITDC - [ITDC (mg CCS)] + [0.25×ITDC (mg ACC)] Subjects will receive instructions regarding the new doses of ACC and will be reminded to take XXX tablets a day, XXX in the morning, XXX in midday and XXX in the evening, before or after a meal (based on their initial assignment). Subjects will be reminded to continue their routine medications consumption during the trial.

Subjects will receive a container to perform 24 hour urine collection prior to their next scheduled visit.

I-Day 27 (±1) by phone: Subjects will be reminded to perform 24 hour urine collection.

I-Day 28 (±1) - Termination of phase I: Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will provide the container of 24 hour urine collection for Ca, P and creatinine to test calciuria. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

Phase I results will be examined before deciding whether or not to embark on the crossover portion of the study planned for Phase II. Phase I data will be summarized, showing for each subject, by arm and overall the relationship between CA levels by amount of ACC replacement of CCS received.

Phase II Ten (10) subjects previously diagnosed and chronically treated for primary hypoparathyroidism will be enrolled. Subjects participated in phase I will be offered to participate in phase II as well. If needed, new subjects will be enrolled.

The subjects will be randomly assigned to one of the following treatments for 6 weeks:

1. Standard of care (CCS) - The same elemental calcium dosage that was used routinely prior to the study.
2. ACC - The established dosage of elemental calcium from ACC (based on the conversion factor and the fed/fasted conditions found in phase I of the study).

The two formulations will be administered with the regular daily dosage of vitamin D (1-alfa D3).

At the end of the treatment, each group will receive the alternative formulation for another 6 weeks.

The superior absorption of ACC will be evaluated using weekly blood tests to calculate serum CA values. Excretion of calcium in urine will be tested at screening and in the end of each treatment.

II-Day -21 (+/-17) Screening: Subjects with a diagnosed primary hypoparathyroidism (see section 4.1 for definitions), and who receiving calcium and vitamin D supplementation at least 1 year prior to the beginning of the study and are without major renal or hepatic disease, will be invited to the Clinical Research Center . At the clinic, subjects will be interviewed, their medical history and their current medication will be documented and they will sign an informed consent form (ICF). Subjects will be referred to perform blood tests for Calcium, P and albumin levels. Calculation of CA will be performed. Subjects will be instructed to perform 24 hour urine collection for Ca, P and creatinine levels. Subjects will be asked to fill out a food and medication diary for 3 consecutive days to evaluate their daily dietary calcium intake. Women of childbearing age will undergo a urine pregnancy test. Eligible subjects, complying with all inclusion criteria and having none of the exclusion criteria will be enrolled to the study.

Subjects will be informed by phone or on site whether they are eligible to enter the study.

II-Day 0: Eligible subjects will arrive at the Clinical Research Center where they will be asked about any changes in their medical condition since their last visit. Blood tests will be performed to define serum calcium, P and albumin baseline values. CA values will be calculated at baseline.

Subjects will be randomly assigned to one of the following treatments:

1. Standard-of-care (CCS) - The same elemental calcium dosage that was used routinely prior to the study.
2. ACC - The established dosage of elemental calcium from ACC (based on the conversion factor and the fed/fasted conditions found in phase I of the study).

Subjects that were assigned to the ACC treatment arm, will receive a pack of ACC tablets, each tablet containing 200 mg elemental calcium (35 day supply + 5 spare tablets). Subjects assigned to the CCS treatment arm will continue to take their routine calcium supplementation.

The exact dosage of calcium supplementation will be determined for each subject according the known medical history.

Subjects will be instructed to continue their routine medications consumption during the trial.

II-Day 3 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). If CA values are within the desired target range (7.0-10.0 mg/dl), subjects will continue to take the calcium doses that were instructed on II-day 0. If CA levels are below 7.0 mg/dL or above 10.0 mg/dL, changes to calcium intake will be made, according to the doctor's decision

II-Day 7 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression). Adjustments of ACC or CCS intake will be performed if necessary.

Subjects will be reminded to take the calcium supplementation according to their assignment instructions.

Subjects will be reminded to continue their routine medications consumption during the trial.

II-Day 10 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). If CA levels are within the desired target range (7.0-10.0 mg/dl), subjects will continue to take the calcium doses that were instructed on II-day 7. If CA levels are below 7.0 mg/dL, or above 10.0 mg/dL, changes to the calcium intake will be made, according to the doctor's decision

II-Day 14 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

Subjects will be reminded to take the calcium supplementation according to their assignment instructions.

Subjects will be reminded to continue their routine medications consumption during the trial.

II-Day 21 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin will be tested. Calculation of CA will be performed. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

Subjects will be reminded to take the calcium supplementation according to the instructions.

Subjects will be reminded to continue their routine medications consumption during the trial.

Subjects will receive a container to perform 24 hour urine collection prior to their next scheduled visit.

II-Day 34 (±1) by phone: Subjects will be reminded to perform 24 hour urine collection.

II-Day 35 (±1): Subjects will arrive to the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will provide the container with 24 hour urine collection for Ca, P and creatinine to test calciuria. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

Subjects previously assigned to the CCS treatment arm will receive a pack of ACC tablets, each tablet containing 200 mg elemental calcium (35 day supply + 5 spare tablets). Subjects previously assigned to the ACC treatment arm, will be instructed to resume their regular CCS supplementation.

The exact dosage of calcium supplementation for each subject will be determined by the known medical history.

Subjects will be reminded to continue their routine medications consumption during the trial.

II-Day 38 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). If CA levels are within the desired target range (7.0-10.0 mg/dl), subjects will continue to take the calcium doses that were instructed on II-day 35. If CA levels are below 7.0 mg/dl or above 10.0 mg/dl, changes to the calcium intake will be made, according to the doctor's decision

II-Day 42 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression). Adjustments of ACC or CCS intake will be performed if necessary.

Subjects will be reminded to take the calcium supplementation according to their assignment instructions.

Subjects will be reminded to continue their routine medications consumption during the trial.

II-Day 45 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed to exclude hypocalcaemia (Ca<7.0 mg/dL). If CA levels are within the desired target range (7.0-10.0 mg/dl), subjects will continue to take the calcium doses that were instructed on II-day 42. If CA levels are below 7.0 mg/dl or above 10.0 mg/dl, changes to the calcium intake will be made, according to the doctor's decision

II-Day 49 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

Subjects will be reminded to take the calcium supplementation according to their assignment instructions.

Subjects will be reminded to continue their routine medications consumption during the trial.

II-Day 56 (±1): Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

Subjects will be reminded to take the calcium supplementation according to their assignment instructions.

Subjects will be reminded to continue their routine medications consumption during the trial.

Subjects will receive a container to perform 24 hour urine collection prior to their next scheduled visit.

II-Day 69 (±1) by phone: Subjects will be reminded to perform 24 hour urine collection.

II-Day 70 (±1) - Termination of phase II: Subjects will arrive at the Clinical Research Center and their serum calcium, P and albumin levels will be tested. Calculation of CA will be performed. Subjects will provide the container with 24 hour urine collection for Ca, P and creatinine to test calciuria. Subjects will be asked about any side effects or AEs that may have occurred and changes in concomitant medications since their last visit. Subjects will be asked about symptoms and signs related with a change in serum calcium levels (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).

ELIGIBILITY:
Inclusion Criteria:

* Primary Hypoparathyroidism - low levels of intact PTH during hypocalcemia at diagnosis.
* Subjects receiving calcium and vitamin D supplementation at least 1 year prior to the beginning of the study.
* Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Subjects who provide written informed consent to participate in the study.
* Age: 18-80, inclusive.

Exclusion Criteria:

* Calcium (albumin corrected) serum values below 7.0 mg/dL or above 10.0 mg/dL
* Any known diseases affecting the absorption from the gastrointestinal tract:

  * Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
  * Chronic diarrhea
* Subjects with neuropsychiatric disease.
* Subjects with impaired renal function (glomerular filtration rate, ≤40 mL/min)
* Subjects with other severe chronic disease requiring long-term therapy.
* Impaired liver function (Liver enzymes> x3 upper limit of normal).
* Subjects with history or presence of kidney stones
* Recurrent urinary tract infections
* Subjects taking drugs which might affect calcium levels such as:

  * Fusid
  * Anticonvulsants
  * Carbonic anhydrase
  * Adrenocorticosteroids
* Subjects who are non-cooperative or unwilling to sign consent form.
* Pregnant or breast-feeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06-25 (Actual)

PRIMARY OUTCOMES:
Calcium (albumin-corrected) serum level - composite value based on multiple measurements | Blood tests will be performed for each subject in each CRC visit from day 0 and onward: Phase I: Day 0, 3, 7, 10, 14, 21, 28. Phase II: Day 0, 3, 7, 10, 14, 21, 35, 38, 42, 45, 49, 56, 70.
  The initial assessment of hypocal¬cemia is usually based on the measurement of serum total calcium corrected for albumin concentration. Normal CA values range from 8.5 to 10.2 mg/dL. In subjects with hypoparathyroidism, the desired target CA values are 7.0-10.0 mg/dL.
  The relationship between total serum calcium and albumin is defined by the following rule: the serum total calcium concentration falls by 0.8 mg/dL for every 1-g/dL fall in serum albumin concentration. This rule assumes that normal albumin equals 4.0 g/dL and normal calcium is 10.0 mg/dL.
  Calculation: Calcium (corrected, mmol/L) = Calcium (measured, mmol/L) + {(40 - albumin(g/L)) x 0.02}

SECONDARY OUTCOMES:
Urine calcium level - 24h urine collection | Phase I: Termination of study (Day 28)
  For a 24-hour urine collection, all of the urine over a 24-hour time period must be collected. The urine sample must include the last urine, 24 hours after starting the collection.
  Urine calcium level > 300 mg/24 hours or > 4 mg/kg of weight/24 hours is considered as hypercalciuria.
Phosphorous serum level - composite value based on multiple measurements | Blood tests will be performed for each subject in each CRC visit from day 0 and onward: Phase I: Day 0, 3, 7, 10, 14, 21, 28. Phase II: Day 0, 3, 7, 10, 14, 21, 35, 38, 42, 45, 49, 56, 70
  The serum phosphorus test measures the amount of phosphate in the blood. Normal values range from 2.4 - 4.1 mg/dL
Urine calcium level - 24h urine collection | Phase II: Day 35
  For a 24-hour urine collection, all of the urine over a 24-hour time period must be collected. The urine sample must include the last urine, 24 hours after starting the collection.
  Urine calcium level > 300 mg/24 hours or > 4 mg/kg of weight/24 hours is considered as hypercalciuria.
Urine calcium level - 24h urine collection | Phase II: termination of study (Day 70)
  For a 24-hour urine collection, all of the urine over a 24-hour time period must be collected. The urine sample must include the last urine, 24 hours after starting the collection.
  Urine calcium level > 300 mg/24 hours or > 4 mg/kg of weight/24 hours is considered as hypercalciuria.
Assessment of symptoms and signs related with hypocalcemia - composite value based on multiple measurements | Phase I: Day 7, 14, 21, 28 Phase II: Day 7, 14, 21, 35, 42, 49, 56, 70
  At each visit to the CRC, subjects will be asked to answer questions for the presence of symptoms and signs related with hypocalcemia (tetany, facial grimacing, paresthesias, muscle aches, arrhythmia, depression).
Urine creatinine level - 24h urine collection | Phase I: Termination of study (Day 28)
  For a 24-hour urine collection, all of the urine over a 24-hour time period must be collected. The urine sample must include the last urine, 24 hours after starting the collection.
  A creatinine clearance test is done on a sample of urine collected over 24 hours. It is used to determine glomerular filtration rate, which helps to measure how well the kidney functions. The normal adult urine calcium/creatinine ratio is <220 mg/g
Urine creatinine level - 24h urine collection | Phase II: Day 35
  For a 24-hour urine collection, all of the urine over a 24-hour time period must be collected. The urine sample must include the last urine, 24 hours after starting the collection.
  A creatinine clearance test is done on a sample of urine collected over 24 hours. It is used to determine glomerular filtration rate, which helps to measure how well the kidney functions. The normal adult urine calcium/creatinine ratio is <220 mg/g
Urine creatinine level - 24h urine collection | Phase II: termination of study (Day 70)
  For a 24-hour urine collection, all of the urine over a 24-hour time period must be collected. The urine sample must include the last urine, 24 hours after starting the collection.
  A creatinine clearance test is done on a sample of urine collected over 24 hours. It is used to determine glomerular filtration rate, which helps to measure how well the kidney functions. The normal adult urine calcium/creatinine ratio is <220 mg/g
Urine phosphorus level - 24h urine collection | Phase I: Termination of study (Day 28)
  The phosphate urine test measures the amount of phosphate in a sample of urine collected over 24 hours (24-hour urine test). Phosphate is a charged ion that contains the mineral phosphorus.
  Results of a test to measure phosphate in urine are seldom useful on their own. They should always be interpreted along with the results of other tests. Calcium and phosphate levels are often measured at the same time.
Urine phosphorus level - 24h urine collection | Phase II: Day 35
  The phosphate urine test measures the amount of phosphate in a sample of urine collected over 24 hours (24-hour urine test). Phosphate is a charged ion that contains the mineral phosphorus.
  Results of a test to measure phosphate in urine are seldom useful on their own. They should always be interpreted along with the results of other tests. Calcium and phosphate levels are often measured at the same time.
Urine phosphorus level - 24h urine collection | Phase II: termination of study (Day 70)
  The phosphate urine test measures the amount of phosphate in a sample of urine collected over 24 hours (24-hour urine test). Phosphate is a charged ion that contains the mineral phosphorus.
  Results of a test to measure phosphate in urine are seldom useful on their own. They should always be interpreted along with the results of other tests. Calcium and phosphate levels are often measured at the same time.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Ish-Shalom, MD, Principal Investigator; Dity Natan, McS, Study Director — Amorphical Ltd.
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Brandi ML, Bilezikian JP, Shoback D, Bouillon R, Clarke BL, Thakker RV, Khan AA, Potts JT Jr. Management of Hypoparathyroidism: Summary Statement and Guidelines. J Clin Endocrinol Metab. 2016 Jun;101(6):2273-83. doi: 10.1210/jc.2015-3907. Epub 2016 Mar 4. PMID 26943719
- [Background] Bilezikian JP, Matsumoto T, Bellido T, Khosla S, Martin J, Recker RR, Heaney R, Seeman E, Papapoulos S, Goldring SR. Targeting bone remodeling for the treatment of osteoporosis: summary of the proceedings of an ASBMR workshop. J Bone Miner Res. 2009 Mar;24(3):373-85. doi: 10.1359/jbmr.090105. No abstract available. PMID 19260805
- [Background] Rubin MR, Dempster DW, Kohler T, Stauber M, Zhou H, Shane E, Nickolas T, Stein E, Sliney J Jr, Silverberg SJ, Bilezikian JP, Muller R. Three dimensional cancellous bone structure in hypoparathyroidism. Bone. 2010 Jan;46(1):190-5. doi: 10.1016/j.bone.2009.09.020. Epub 2009 Sep 25. PMID 19782782
- [Background] Fong J, Khan A. Hypocalcemia: updates in diagnosis and management for primary care. Can Fam Physician. 2012 Feb;58(2):158-62. PMID 22439169
- [Background] Cusano NE, Rubin MR, Sliney J Jr, Bilezikian JP. Mini-review: new therapeutic options in hypoparathyroidism. Endocrine. 2012 Jun;41(3):410-4. doi: 10.1007/s12020-012-9618-y. Epub 2012 Feb 7. PMID 22311174
- [Background] Straub DA. Calcium supplementation in clinical practice: a review of forms, doses, and indications. Nutr Clin Pract. 2007 Jun;22(3):286-96. doi: 10.1177/0115426507022003286. PMID 17507729
- [Background] Bilezikian JP, Cusano NE, Khan AA, Liu JM, Marcocci C, Bandeira F. Primary hyperparathyroidism. Nat Rev Dis Primers. 2016 May 19;2:16033. doi: 10.1038/nrdp.2016.33. PMID 27194212